CLINICAL TRIAL: NCT07064720
Title: Adding Dexmedetomidine to Mannitol to Attenuate the Increase of Intracranial Pressure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Assistant Professor of anesthesia, SICU & and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-50-2024
Record Dates: First submitted 2025-07-06; First posted 2025-07-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Dexmedetomidine
Keywords: dexmedetomidine; mannitol
MeSH Terms: interventions — Dexmedetomidine; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (D) (Experimental): Dexmedetomidine with Mannitol
  Interventions: Drug: Dexmedetomidine with Mannitol
- Group (M) (Experimental): Mannitol only
  Interventions: Drug: Mannitol (20%)

INTERVENTIONS:
Drug: Dexmedetomidine with Mannitol — receive 1 mcg/kg of dexmedetomidine added to 0.4 mcg/kg of mannitol
  Arms: Group (D)
Drug: Mannitol (20%) — receive 0.5 g/kg of mannitol
  Arms: Group (M)

SUMMARY:
Dexmedetomidine is a potent alpha-2 adrenergic receptor agonist. In addition, dexmedetomidine-induced stimulation of the postsynaptic alpha-2 adrenergic receptor on the cerebral blood vessels can cause cerebral vasoconstriction and decrease cerebral blood flow

ELIGIBILITY:
Inclusion Criteria:

ASA I-II Patients scheduled for elective robot-assisted laparoscopic prostatectomy

Exclusion Criteria:

* • ASA physical status > II

  * Cardiac patients
  * Cerebrovascular disease
  * Glaucoma
  * Hepatic failure
  * Renal failure
  * History of anaphylactic reaction to dexmedetomidine or mannitol
  * Hemodynamic instability
  * Cannot measure ONSD for example due to ophthalmological problems.
  * Any cause of preoperative increase in ICP for example intracranial space occupying lesions.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter | 90 minutes

SECONDARY OUTCOMES:
Postoperative neurologic complications | 24 HOURS
Postoperative cardiac complications | 24 hours
Duration of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- facility of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided